CLINICAL TRIAL: NCT06657560
Title: Pharmacokinetics (PK) Study of HRS-9231 Injection in Chinese Subjects With Renal Impairment and Normal Renal Function
Brief Title: Pharmacokinetics, Dialysability and Safety of HRS-9231 in Healthy Volunteers and in Patients With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HRS-9231-103
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Contrast-Enhanced Magnetic Resonance Imaging Detection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A (Experimental): Healthy volunteer with stable normal renal function defined with an absolute value of eGFR ≥ 90 and < 130 mL/min based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 25% between the 2 measurements.
  Interventions: Drug: HRS-9231
- Cohort B (Experimental): Patient with stable mild renal impairment defined with an absolute value of eGFR ≥ 60 and <90 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 25% between the 2 measurements.
  Interventions: Drug: HRS-9231
- Cohort C (Experimental): Patient with stable moderate renal impairment defined with an absolute value of eGFR between ≥ 30 and <60 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements.
  Interventions: Drug: HRS-9231
- Cohort D (Experimental): Patient with stable severe renal impairment defined with an absolute value of eGFR between ≥ 15 and <30 mL/min included based on two eGFR assessments done at screening and inclusion, with a maximum tolerance of 15% between the 2 measurements.
  Interventions: Drug: HRS-9231
- Cohort E (Experimental): Patient with end-stage renal failure who requires 3 hemodialysis sessions per week and defined with an absolute value of eGFR <15 mL/min.
  Interventions: Drug: HRS-9231

INTERVENTIONS:
Drug: HRS-9231 — HRS-9231

SUMMARY:
This is an open-label, non-randomized, parallel cohorts design, multicenter, single dose phase I study.

The primary objectives are:

To evaluate the pharmacokinetics (plasma and urine) profile of HRS-9231 following single intravenous injection (0.05 mmol/kg body weight) in patients with mild to severe renal impairment and in healthy volunteers with normal renal function used as reference.

To assess dialysability of HRS-923 following a single intravenous injection (0.05 mmol/kg body weight) in patients with end stage renal disease requiring hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ages 18 to 65, inclusive, at the time of informed consent.
2. Female subjects weigh ≥ 45 kg, male subjects weigh ≥ 50 kg, and BMI between 18.0 and 28.0 kg/m2, inclusive, at screening.
3. Have an eGFR expressed in mL/min/1.73m2 (MDRD formula estimation) at screening within the range of:

   Cohort A - normal renal function: ≥ 90 mL/min and < 130 mL/min; Cohort B - mild renal impairment: 60 < 90 mL/min; Cohort C - moderate renal impairment: 30 < 60 mL/min; Cohort D - severe renal impairment: 15 < 30 mL/min; Cohort E - ESRD subjects requiring HD: < 15 mL/min.
4. The renal function is required to be stable. The interval between two assessments during the screening period should be at least 72 hours apart (the first renal function assessment result may use historical values with 30 days before screening), and the two assessments should be consistent with the same renal function classification and two values have to show ≤25%. If the two assessments are inconsistent in terms of renal function category, the third assessment has to be conducted at least 72 hours after the second assessment. If the second and third assessments differ, the subject will be ineligible for the study.

Exclusion Criteria:

1. Subject with any history of severe allergic or anaphylactic reactions to any allergen including drugs and contrast agents, or allergic disease diagnosed and treated by a physician.
2. Subject has positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or treponema pallidum antibody.
3. Subjects who have undergone major surgery within 3 months before screening, or those who have received surgery that may significantly affect the pharmacokinetics or safety evaluation of the study drug, are judged by the investigators to be unsuitable for participation.
4. Participated in other clinical trials within 3 months before screening or plan to participate in other clinical trials during this study.
5. Blood loss or blood donation of more than 200 mL within 3 months before screening, or intended to donate blood during or within 1 month after the end of the trial.
6. Those who have been vaccinated with inactivated/live/attenuated vaccines within 1 month before screening or who have an intention to vaccinate during the trial.
7. History of kidney transplantation surgery.
8. Patients with mild, moderate, or severe renal impairment are expected to receive any type of dialysis during the study (cohort B-D); Those who need treatment other than intermittent hemodialysis therapy during the study period, or those who have not been able to maintain a stable hemodialysis of 2 to 4 times per week for at least 1 month before administration (Group E).
9. Incontinence or anuria (e.g., <100 mL/d) in patients with mild, moderate, and severe renal impairment (B-D group).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Cmax | Prior to HRS-9231 administration and Day 5 (for all cohorts) or Day 6 (only for cohort D).
  Observed maximum plasma concentration. Blood samples will be collected.
AUC0-t | Prior to HRS-9231 administration and Day 5 (for all cohorts) or Day 6 (only for cohort D).
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected.
AUC0-∞ | Prior to HRS-9231 administration and Day 5 (for all cohorts) or Day 6 (only for cohort D).
  Area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected.
Tmax | Prior to HRS-9231 administration and Day 5 (for all cohorts) or Day 6 (only for cohort D).
  Observed time to reach C(max). Blood samples will be collected.
Ae | Prior to HRS-9231 administration and Day 5 (for all cohorts) or within 6 days (only for cohort D) after administration.
  Amount excreted. Urine samples will be collected.

SECONDARY OUTCOMES:
Incidence of treatment emergent AEs (TEAEs) | From screening visit to 6 months after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University First Affiliated Hospital (Shandong Qianfoshan Hospital), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided